CLINICAL TRIAL: NCT05551806
Title: Effectiveness of Internet-based Self-help Cognitive Behavioural Therapy (CBT-I) in Reducing Insomnia Symptoms Among the Adult Population: A Randomized Controlled Trial
Brief Title: Effectiveness of Internet-based Self-help Cognitive Behavioural Therapy in Reducing Insomnia Among Adult Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: Baptist Oi Kwan Social Service (Other)
Responsible Party: Principal Investigator, CHAN Ka Shing Kevin, Associate Professor, Head of Department of Psychology, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-2022-0340
Record Dates: First submitted 2022-09-01; First posted 2022-09-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Insomnia
Keywords: Cognitive Behavioural Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I group (Experimental): Participants in the CBT-I condition start the 6-week CBT-I immediately after randomization, complete the post-intervention assessment right after they finish the treatment, and complete the follow-up assessment 4 weeks after the post-intervention assessment. They will be invited to participate in an interview after completing the post-intervention assessment.
  Interventions: Behavioral: Internet-based self-help cognitive behavioural therapy
- Waitlist control group (No Intervention): Participants in the waitlist control group will wait for 6 weeks without the CBT-I intervention and then complete the post-intervention assessment; while waiting for 4 more weeks and then completing the follow-up assessment. The waitlist control participants will start CBT-I (equivalent to that of the CBT-I group) immediately after completing the follow-up assessment.

INTERVENTIONS:
Behavioral: Internet-based self-help cognitive behavioural therapy — The online CBT-I course will consist of an introductory module, followed by 6 weekly modules, incorporating the key CBT-I components, including sleep hygiene education, stimulus control, sleep restriction, relaxation training, and cognitive therapy.
  Arms: CBT-I group

SUMMARY:
This experimental study aims to develop an internet-based self-help cognitive behavioural therapy for insomnia that reduces insomnia symptoms and its associated adverse outcomes among people with sub-threshold insomnia symptoms. In particular, this study compares the efficacy of internet-delivered self-help CBT-I with the wait-list control group, in treating insomnia in a non-clinical population.

The online CBT-I course will consist of an introductory module, followed by 6 weekly modules. Each module will consist of the main treatment component presented in written or video format, quiz, and homework. Materials will be presented in an interactive manner to facilitate engagement.

DETAILED DESCRIPTION:
Although the Internet self-help CRT-I program have shown promising effect on dealing with insomnia symptoms, the effectiveness of internet self-help CBT-I in adults with sub-clinical insomnia symptoms in Hong Kong is under-studied. Therefore, the present study aimed to compare the efficacy of internet-delivered self-help CBT-I with the wait-list control group, in treating insomnia in a non-clinical population. We hypothesized that (1) participants who received CBT-I treatment would have improved insomnia symptoms after the intervention as compared with the wait-list controls; (2) participants from CBT-I would have better sleep hygiene, and less dysfunctional beliefs about sleep and pre-sleep arousal after the intervention as compared with the wait-list controls; (3) participants from CBT-I would have improved mental health, daytime functioning, quality of life, and general well-being after treatment, as compared with the wait-list controls.

The online CBT-I course will consist of an introductory module, followed by 6 weekly modules, incorporating the key CBT-I components, including sleep hygiene education, stimulus control, sleep restriction, relaxation training, and cognitive therapy. Each module will consist of the main treatment component presented in written or video format, quiz, and homework. Materials will be presented in an interactive manner to facilitate engagement.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents
* Age ≥18 years
* Insomnia Severity Index score > 7 and < 22
* Being able to read Chinese
* Have a computer, tablet and/or smartphone device with Internet access
* have a regular email address
* Willing to give informed consent and comply with the trial protocol

Exclusion Criteria:

* Receiving psychological treatment at least once per month
* Currently taking prescribed psychiatric drugs such as antidepressants, tranquilizers, and sleeping pills regularly
* Carrying a diagnosis of psychosis or schizophrenia
* Participating in any other academic studies or clinical trials related to insomnia
* Having current suicidal plans or acts or having had suicidal plans or acts within the past 12 months
* Shift workers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Assessment in the Severity of Sleep Problem on the Insomnia Severity Index (ISI) at Post-Intervention Assessment and Follow-up Assessment | Before intervention, Immediately after intervention, and 4 weeks after intervention
  The ISI assesses the change in a 5-point Likert scale, ranging from 1 (none/ very dissatisfied/ not at all noticeable, worried & interfering) to 5 (very severe/ very satisfied/ very much noticeable, worried & interfering).

SECONDARY OUTCOMES:
Change from Baseline Assessment in General Sleep Disturbances on the Pittsburgh Sleep Quality Index (PSQI) at Post-Intervention Assessment and Follow-up Assessment | Before intervention, Immediately after intervention, and 4 weeks after intervention
  The PSQI assesses the change in a 4-point Likert scale, ranging from 1 (not during the past month/ very good) to 4 (three or more times a week/ very poor).
Change from Baseline Assessment in Daily Sleep-Wake Schedule on the 7-Day Consensus Sleep Diary at Post-Intervention Assessment and Follow-up Assessment | Before intervention, Immediately after intervention, and 4 weeks after intervention
  The 7-day consensus sleep diary will calculate the change of participants' sleep parameters from the diary data.
Change from Baseline Assessment in Cognitive and Somatic Manifestations of Arousal on the Pre-sleep Arousal Scale (PSAS) at Post-Intervention Assessment and Follow-up Assessment | Before intervention, Immediately after intervention, and 4 weeks after intervention
  The PSAS assesses the change in a 5-point Likert scale, ranging from 1 (not at all) to 5 (extremely).
Change from Baseline Assessment in Sleep Habits on the Sleep Hygiene Practice Scale (SHPS) at Post-Intervention Assessment and Follow-up Assessment | Before intervention, Immediately after intervention, and 4 weeks after intervention
  The SHPS assesses the change in a 6-point Likert scale, ranging from 1 (never) to 6 (always).
Change from Baseline Assessment in Sleep Related Cognition on the Dysfunctional Beliefs and Attitudes about Sleep (DBAS) at Post-Intervention Assessment and Follow-up Assessment | Before intervention, Immediately after intervention, and 4 weeks after intervention
  The DBAS assesses the change in a 10-point Likert scale, ranging from 0 (strongly disagree) to 10 (strongly agree).
Change from Baseline Assessment in Psychological Wellbeing on the World Health Organisation-Five Well-Being Index (WHO-5) at Post-Intervention Assessment and Follow-up Assessment | Before intervention, Immediately after intervention, and 4 weeks after intervention
  The WHO-5 assesses the change in a 6-point Likert scale, ranging from 1 (never) to 6 (all of the time).
Change from Baseline Assessment in Psychological Distress on the Short Form of the Depression, Anxiety, and Stress Scale (DASS-21) at Post-Intervention Assessment and Follow-up Assessment | Before intervention, Immediately after intervention, and 4 weeks after intervention
  The DASS-21 assesses the change in a 4-point Likert scale, ranging from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time).
Change from Baseline Assessment in Quality of Life on the Twelve-Item Short-Form (SF-12) Health Survey at Post-Intervention Assessment and Follow-up Assessment | Before intervention, Immediately after intervention, and 4 weeks after intervention
  The SF-12 assesses the change in a combination of 5-point and 3-point Likert scale, ranging respectively from 1 (poor/ never) to 5 (excellent/ very much), and 1 (never) to 3 (very much).
Change from Baseline Assessment in Functional Impairment of Insomnia on the Work and Social Adjustment Scale (WSAS) at Post-Intervention Assessment and Follow-up Assessment | Before intervention, Immediately after intervention, and 4 weeks after intervention
  The WSAS assesses the change in a 9-point Likert scale, ranging from 1 (not at all) to 9 (very severely).
Change from Baseline Assessment in Cognitive Failure on the Measure of Insight into Cognition-Self Report (MIC-SR) at Post-Intervention Assessment and Follow-up Assessment | Before intervention, Immediately after intervention, and 4 weeks after intervention
  The MIC-SR assesses the change in a 4-point Likert scale, ranging from 1 (never) to 4 (almost daily).
Change from Baseline Assessment in Expectation toward Intervention on the Credibility of Treatment Rating Scale (CTRS) at Post-Intervention Assessment and Follow-up Assessment | Before intervention, Immediately after intervention, and 4 weeks after intervention
  The CTRS assesses the change in a 6-point Likert scale, ranging from 1 (not at all confident) to 6 (very confident).
Insomnia Treatment Acceptability assessed the Insomnia Treatment Acceptability Scale (ITAS) at the Interview after Post-Intervention Assessment | Immediately after Post-Intervention Assessment
  The ITAS assesses the insomnia treatment acceptability in a 10-point Likert scale, ranging from 1 (not at all acceptable) to 10 (very acceptable).
Treatment Adherence at the Interview after Post-Intervention Assessment | Immediately after Post-Intervention Assessment
  Participants report the number of sessions they had read, how long they had spent on the CBT program, and how far they had followed the instructions.
Treatment Satisfaction at the Interview after Post-Intervention Assessment | Immediately after Post-Intervention Assessment
  Participants report on whether they like, found it useful, and improvement of the intervention in a 10-point Likert scale, ranging from 0 (not at all suitable) to 10 (very suitable).
Treatment Satisfaction in internet (Acceptability of the Internet for delivering CBT) at the Interview after Post-Intervention Assessment | Immediately after Post-Intervention Assessment
  Participants report on how suitable, how convenient, how much they liked, and how worried they were about their privacy in a 10-point Likert scale, ranging from 0 (not at all suitable) to 10 (very suitable).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin, Ka Shing CHAN, Principal Investigator — The Education University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Baptist Oi Kwan Social Service, Hong Kong
  - The Education University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT05551806/ICF_000.pdf